CLINICAL TRIAL: NCT02739698
Title: Role of Intraperitoneal Intraoperative Chemotherapy With Paclitaxel in the Surgical Treatment of Peritoneal Carcinomatosis From Ovarian Cancer. Hyperthermia Versus Normothermia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Principal Investigator, Sebastián Rufián, PhD, MD, Maimónides Biomedical Research Institute of Córdoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI 0678-10
Record Dates: First submitted 2016-04-04; First posted 2016-04-15 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Peritoneal Carcinomatosis
Keywords: ovarian cancer
MeSH Terms: conditions — Peritoneal Neoplasms; Ovarian Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- normothermic (36-37ºC) (Experimental): Group 1, n=16(normothermic): Intraperitoneal administration of 60 mg/m2 paclitaxel per 2 liters of 1.5% dextrose in room temperature (36-37ºC).
  Interventions: Drug: Paclitaxel; Procedure: Radical surgery-peritonectomy
- hyperthermic (41-42ºC) (Experimental): Group 2, n=16 (hyperthermic): Intraperitoneal administration of 60 mg/m2 paclitaxel per 2 liters of 1.5% dextrose in continuous hyperthermic perfusion (41-42ºC).
  Interventions: Drug: Paclitaxel; Procedure: Radical surgery-peritonectomy

INTERVENTIONS:
Drug: Paclitaxel
Procedure: Radical surgery-peritonectomy

SUMMARY:
A randomized controlled single-blind clinical trial was performed, in 32 patients diagnosed with peritoneal carcinomatosis from epithelial ovarian cancer, who underwent radical surgery-peritonectomy, achieving an optimal R0-R1 cytoreduction (microscopic tumor residues (R0) or macroscopic tumor residues < 1cm (R1)) followed by hyperthermia against normothermia intraperitoneal intraoperative chemotherapy with paclitaxel

ELIGIBILITY:
Inclusion Criteria:

1. age ranged between 18 and 75 years old;
2. histopathologic confirmation of peritoneal carcinomatosis from epithelial ovarian cancer (stage IIIc- FIGO (International Federation of Gynecology and Obstetrics));
3. Karnofsky index > 70 or performance status ≤2;
4. informed consent form filled out correctly.

Exclusion Criteria:

1. unfulfillment of inclusion criteria;
2. extraabdominal metastasis or stage IV FIGO (liver, lung, bone, etc);
3. concomitance of another malignant neoplasm;
4. renal, hepatic or cardiovascular dysfunction;
5. intolerance during the treatment; - (6) refusal to participate in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2017-03 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fernandez-Peralbo MA, Priego-Capote F, Luque de Castro MD, Casado-Adam A, Arjona-Sanchez A, Munoz-Casares FC. LC-MS/MS quantitative analysis of paclitaxel and its major metabolites in serum, plasma and tissue from women with ovarian cancer after intraperitoneal chemotherapy. J Pharm Biomed Anal. 2014 Mar;91:131-7. doi: 10.1016/j.jpba.2013.12.028. Epub 2014 Jan 2. PMID 24447964

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 43 subjects were recruited but 11 were excluded after the pathologist samples review
Groups:
- Normothermic (36-37ºC): Group 1, n=16(normothermic): Intraperitoneal administration of 60 mg/m2 paclitaxel per 2 liters of 1,5% dextrose in room temperature (36-37ºC).
  Paclitaxel
  Radical surgery-peritonectomy (ovarian carcinomatosis)
- Hyperthermic (41-42ºC): Group 2, n=16 (hyperthermic): Intraperitoneal administration of 60 mg/m2 paclitaxel per 2 liters of 1,5% dextrose in continuous hyperthermic perfusion (41-42ºC).
  Paclitaxel
  Radical surgery-peritonectomy (ovarian carcinomatosis)
Period: Overall Study
Arm/Group | Normothermic (36-37ºC) | Hyperthermic (41-42ºC)
Started | 22 | 21
Completed | 16 | 16
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normothermic (36-37ºC) | Hyperthermic (41-42ºC) | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 4 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Grouped Miller and Payne (MP) System for Pathological Response: G1 (Minimal Changes and < 30% Cells Tumour Reduction That Includes MP G1-G2), G3 (Microscopic Foci, Cells Tumour Reduction up to >90% That Includes MP G3-G4) and G5 (no Residual Tumour)
Description: Histopathology scoring system to assess response, previous and post intraperitoneal intraoperative chemotherapy. Compare cancer cellularity of the biopsy (before treatment) with the other biopsy (after treatment).
Time Frame: The biopsies were taken before and after the treatment (intraperitoneal intraoperative chemotherapy for 60 minutes) and then they were analysed by two blinded pathologists.
Measure: Number; unit: percentage of complete pathological resp
Groups:
- Normothermic (36-37ºC): Group 1, n=16(normothermic): Intraperitoneal administration of 60 mg/m2 paclitaxel per 2 liters of 1,5% dextrose in room temperature (36-37ºC).
  Paclitaxel
  Radical surgery-peritonectomy
- Hyperthermic (41-42ºC): Group 2, n=16 (hyperthermic): Intraperitoneal administration of 60 mg/m2 paclitaxel per 2 liters of 1,5% dextrose in continuous hyperthermic perfusion (41-42ºC).
  Paclitaxel
  Radical surgery-peritonectomy
Arm/Group | Normothermic (36-37ºC) | Hyperthermic (41-42ºC)
Number analyzed (Participants) | 16 | 16
percentage of complete pathological resp | 18.8 | 25

ADVERSE EVENTS:
Arm/Group | Normothermic (36-37ºC) | Hyperthermic (41-42ºC)
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No